CLINICAL TRIAL: NCT03319771
Title: Effects of Exercise Training on Learning and Memory Outcomes in Multiple Sclerosis
Brief Title: Exercise and Learning and Memory in Multiple Sclerosis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Termination of study funding due to COVID-19
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: EMD Serono (Industry)
Responsible Party: Principal Investigator, Brian Sandroff, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 300000373
Record Dates: First submitted 2017-10-13; First posted 2017-10-24 (Actual); Last update posted 2021-10-11 (Actual); Status verified 2021-10

CONDITIONS: Multiple Sclerosis; Physical Activity; Memory Impairment; Cognitive Change
Keywords: exercise; neuroimaging; walking; multiple sclerosis
MeSH Terms: conditions — Multiple Sclerosis; Motor Activity; Memory Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treadmill Walking Exercise Training (Experimental): 12 weeks of supervised, progressive treadmill walking exercise training
  Interventions: Behavioral: Treadmill Walking Exercise Training
- Stretching-and-toning Exercise Training (Active Comparator): 12 weeks of supervised, stretching-and-toning exercise training
  Interventions: Behavioral: Stretching-and-toning Exercise Training

INTERVENTIONS:
Behavioral: Treadmill Walking Exercise Training — 12-weeks of supervised, progressive treadmill walking exercise training
  Arms: Treadmill Walking Exercise Training
Behavioral: Stretching-and-toning Exercise Training — 12-weeks of supervised, stretching-and-toning exercise training
  Arms: Stretching-and-toning Exercise Training

SUMMARY:
The two primary study objectives involve examining the effects of treadmill walking exercise training versus stretching-and-toning activities on the primary and secondary outcomes.

Specific Aim 1: The first specific aim is to examine the effects of 3-months of treadmill walking exercise training compared with an active control condition on learning and memory outcomes in fully-ambulatory persons with MS who have impairment in learning new information. We hypothesize that those who undergo treadmill walking exercise training will demonstrate improvements in learning and memory relative to those who undergo stretching-and-toning activities.

Specific Aim 2: The second specific aim is to examine the effects of 3-months of treadmill walking exercise training compared with an active control condition on hippocampal volume, hippocampal resting-state functional connectivity, and cardiorespiratory fitness in those persons with MS. We hypothesize that those who are randomly assigned to the treadmill walking exercise condition will demonstrate increases in hippocampal volume and resting-state functional connectivity (i.e., adaptive increases) and improved cardiorespiratory fitness relative to those in the stretching-and-toning condition.

DETAILED DESCRIPTION:
The proposed study involves a single-blind, Phase I randomized controlled trial (RCT) on the effects of supervised treadmill walking exercise training on learning and memory, hippocampal structure/function, and cardiorespiratory fitness outcomes in fully-ambulatory (i.e., EDSS ≤ 4.0) persons with multiple sclerosis (MS) who have impairment in learning new information. This study will compare the effects of 3 months of supervised, progressive (both intensity and duration) chronic treadmill walking exercise (designed based on pilot work [Sandroff et al., 2015; 2016a; 2016b] and American College of Sports Medicine (ACSM) guidelines) with those of an active control condition (i.e., stretching-and-toning activities) on learning and memory, hippocampal volume and resting-state functional connectivity, and cardiorespiratory fitness. Learning and memory represents the primary outcome, whereas hippocampal volume and resting-state functional connectivity and cardiorespiratory fitness represent the secondary outcomes. Such an investigation will provide the first Class I evidence for the effects of treadmill walking exercise training on those outcomes in MS.

During baseline, participants will first complete a battery of neuropsychological tests, followed by an incremental exercise test to exhaustion on a motor-driven treadmill to measure cardiorespiratory fitness, and will undergo a MRI scan. Those outcomes will be measured by assessors who are blinded to condition. Participants will undertake several neuropsychological tests addressing various aspects of learning and memory. These tests include the California Verbal Learning Test-2 [Delis et al., 2000] and Selective Reminding Task [Buschke & Fuld, 1974] as measures of verbal learning and memory, and the Brief Visuospatial Memory Test-Revised [Benedict, 1997] and 10/36 Spatial Recall Test [Rao et al., 1984] as measures of visuospatial learning and memory. Cognitive processing speed will be measured using the Symbol Digit Modalities Test [Smith, 1982], verbal fluency will be measured using the Controlled Oral Word Association Test [Benton, 1994], and executive control (i.e., inhibitory control) will be measured using a modified flanker task [Eriksen & Eriksen, 1974]. Cardiorespiratory fitness will be measured as peak oxygen consumption (VO2peak), using an incremental exercise test to exhaustion on a motor-driven treadmill and an open-circuit spirometry system (ParvoMedics True One 2400, Sandy, UT) for analyzing expired gases using a modified Balke protocol. This protocol is commonly used for measuring cardiorespiratory fitness in older adults [e.g. Colcombe et al., 2004] and persons with chronic stroke [e.g., Macko et al., 1997] and further is consistent with the ACSM guidelines for exercise testing of MS patients [ACSM, 2013]. Lastly, participants will undergo structural and resting-state functional connectivity magnetic resonance images of the hippocampus. The MR instrument that will be used is an FDA-approved Siemens 3 T clinical imager. Following baseline testing, participants will be randomly assigned to either the exercise training or active control condition using concealment. Participants further will blinded to condition (i.e., unaware that the treadmill walking exercise training condition represents the experimental condition and the stretching-and-toning condition represents the active control condition).

The exercise training will include 3-months of supervised, progressive light, moderate, and vigorous intensity treadmill walking exercise, and will be based on ACSM guidelines for exercise prescription [ACSM, 2013]. We selected treadmill walking exercise as the aerobic exercise modality based on pilot work that suggests that treadmill walking might exert larger beneficial effects on cognition compared with stationary cycling [Sandroff et al., 2015], and that such benefits occur for light, moderate, and vigorous intensity treadmill walking exercise [Sandroff et al., 2016]. The exercise training itself will take place 3 times per week over 3 months, led by trained exercise leaders, and will initially consist of 15 minutes of light-to-moderate intensity treadmill walking exercise and eventually progress to 40 minutes of vigorous intensity exercise by month 3. The stretching-and-toning activities will be included as a minimal exercise, active control condition. The control condition will be delivered using the same frequency and duration of the treadmill walking exercise condition. The stretching-and-toning activities will be based on a manual provided by the National Multiple Sclerosis Society, and stretching-and-toning activities will be progressively included over the course of the 3-month study period. Participants will further be asked to not undertake additional exercise (i.e., not join a gym and begin exercising) over the duration of the study. The cognitive, cardiorespiratory fitness, and MRI outcomes will be assessed again following the 3-month study period by assessors who are blinded to condition.

The data will be analyzed using mixed-factor ANOVA with time (pre- and post-) as a within-subjects factor and condition (exercise or control) as a between-subjects factor on learning and memory, hippocampal, and cardiorespiratory fitness outcomes (see Specific Aims/Hypotheses 1 and 2 in the Primary Study Objectives and Study Hypothesis sections). Effect sizes will be expressed as partial eta-squared (ηp2) and Cohen's d [Cohen, 1988]. Spearman's rho rank-order correlations (ρ) will be performed for the associations among changes in cardiorespiratory fitness, hippocampal structure/function, and learning and memory for those who underwent the treadmill walking exercise training condition (See Specific Aims/Hypotheses 3 and 4 in the Secondary Study Objectives and Study Hypothesis sections). The effect sizes from the interaction terms from the ANOVAs and correlations will serve as effect sizes for the subsequent power analyses required for a subsequent Phase II RCT.

ELIGIBILITY:
Inclusion/Exclusion Criteria:

- All participants will:

* Be between the ages of 18-54 (Males 18-44; Females 18-54)
* Have a clinically definite MS diagnosis based on established criteria
* Be fully-ambulatory based on Expanded Disability Status Scale (EDSS) scores between 0-4.0
* Demonstrate impairment in learning new information based on open-trial Selective Reminding Task scores at least 1.5 SD's below the normative score for healthy controls (i.e., 5th percentile)
* Be relapse-free and will not have acutely taken corticosteroids for at least 30 days (i.e., relative neurologic stability)
* Not have a history of major depressive disorder, schizophrenia, bipolar disorder I or II, or substance-abuse disorders.
* Not be taking medications that can affect cognition (e.g., antipsychotics, benzodiazepines).
* Be right-handed
* Have corrected vision better than 20/80
* Not have known/diagnosed cardiovascular, metabolic, or renal disease. Individuals with known/diagnosed cardiovascular, metabolic, or renal disease who are asymptomatic will be included only with a physician's approval.
* Demonstrate scores on the Mini-Mental State Examination (MMSE) of 21 or higher (no decisional impairment)
* Be on a stable disease-modifying therapy regimen (i.e., at least 6 months prior to study enrollment).
* Have a low risk for contraindications for MRI based on not having metal (e.g., non-MRI compatible aneurysm clips, metal shards in the body or eyes, or recently placed surgical hardware) or electronic devices (e.g., pacemaker, cochlear implant) within the body.
* Not be pregnant
* Not be engaging in ≥ 150 min of moderate-to-vigorous physical activity (i.e., not meeting public health guidelines for physical activity) per week
* Not be actively engaging in cognitive rehabilitation, or participating in regular brain fitness activities
* Demonstrate systolic blood pressure values of < 200 mmHg or diastolic blood pressure values < 110 mmHg at rest

Ages: 18 Years to 54 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2020-03-16 (Actual); Study Completion 2021-01-03 (Actual)

PRIMARY OUTCOMES:
Composite Learning and Memory Performance | Baseline to 12-week follow-up
  Composite z-score of performance on California Verbal Learning Test-II, Selective Reminding Task, Brief Visuospatial Memory Test-Revised, and 10/36 Spatial Recall Test

SECONDARY OUTCOMES:
Hippocampal Volume | Baseline to 12-week follow-up
  Volume of bilateral hippocampi measured using structural MRI

CONTACTS AND LOCATIONS:
Overall Officials: Brian M Sandroff, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sandroff BM, Wylie GR, Baird JF, Jones CD, Diggs MD, Genova H, Bamman MM, Cutter GR, DeLuca J, Motl RW. Effects of walking exercise training on learning and memory and hippocampal neuroimaging outcomes in MS: A targeted, pilot randomized controlled trial. Contemp Clin Trials. 2021 Nov;110:106563. doi: 10.1016/j.cct.2021.106563. Epub 2021 Sep 5. PMID 34496278
- [Derived] Sandroff BM, Motl RW, Bamman M, Cutter GR, Bolding M, Rinker JR, Wylie GR, Genova H, DeLuca J. Rationale and design of a single-blind, randomised controlled trial of exercise training for managing learning and memory impairment in persons with multiple sclerosis. BMJ Open. 2018 Dec 14;8(12):e023231. doi: 10.1136/bmjopen-2018-023231. PMID 30552263